CLINICAL TRIAL: NCT00686699
Title: A Phase 2a, Multiple Dose, Placebo Controlled, Randomized, Two Way Crossover Study to Assess the Efficacy of SCH 420814 in Reducing Anti Psychotic-Induced Extra Pyramidal Symptoms Among Subjects With Schizophrenia and Schizoaffective Disorders
Brief Title: Study of Preladenant for the Treatment of Antipsychotic Induced Movement Disorders in Participants With Schizophrenia (Study P04628)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated after 9 participants completed due to lack of enrollment for 6 months.
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P04628; 2005-006048-42 (EudraCT Number); MK-3814-014 (Other: Merck Protocol Number)
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Results first posted 2016-12-07 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-10

CONDITIONS: Akathisia, Drug-Induced; Dyskinesia, Drug-Induced; Parkinsonian Disorders
Keywords: Anti-Dyskinesia Agents; Antipsychotic Agents
MeSH Terms: conditions — Akathisia, Drug-Induced; Dyskinesia, Drug-Induced; Parkinsonian Disorders | interventions — 2-(2-furanyl)-7-(2-(4-(4-(2-methoxyethoxy)phenyl)-1-piperazinyl)ethyl)-7H-pyrazolo(4,3-e)(1,2,4)triazolo(1,5-c)pyrimidine-5-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preladenant 25 mg BID→Placebo BID (Experimental): Participants received one preladenant 25 mg capsule twice daily (BID) for 14 days during the first treatment period and received one matching placebo capsule BID during the second treatment period. The 2 treatment periods were separated by a 3-week washout period.
  Interventions: Drug: Preladenant
- Placebo BID→Preladenant 25 mg BID (Placebo Comparator): Participants received one matching placebo capsule BID for 14 days during the first treatment period and received one preladenant 25 mg capsule during the second treatment period. The 2 treatment periods were separated by a 3-week washout period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Preladenant — capsules
  Other Names: SCH 420814; MK-3814
  Arms: Preladenant 25 mg BID→Placebo BID
Drug: Placebo — capsules
  Arms: Placebo BID→Preladenant 25 mg BID

SUMMARY:
This study was designed to determine if preladenant (SCH 420814, MK-3814) can reduce drug-induced involuntary movements in participants with schizophrenia or schizoaffective disorder. Participants were to be evaluated for two 14-day treatment periods with a 3-week washout period between treatment periods. The primary outcome measure, Extrapyramidal Symptom Rating Score (ESRS), was to be evaluated frequently during the treatment periods.

ELIGIBILITY:
Inclusion Criteria:

* Males or females >=18 and <=65 years old with a body mass index of 17-31 kg/m^2.
* Diagnosed with Diagnostic and Statistical Manual of Mental Disorders, 4th Ed. (DSM-IV) criteria for schizophrenia/schizoaffective (depressive type) disorder with antipsychotic-induced extrapyramidal symptoms (parkinsonism, akathisia, dystonia, or tardive dyskinesia [TD]) based on the following ESRS criteria:

  * parkinsonism, dystonia, or TD - ESRS score >=2 on 2 items or >=3 on one item,
  * akathisia - ESRS score >=3 on two items,
* Has total ESRS score >8.
* Must be receiving neuroleptics at a stable dosage for at least 7 days prior to enrollment.
* Clinical laboratory tests, physical exam, and electrocardiogram must be within normal limits or clinically acceptable to the investigator/sponsor (except signs and symptoms of Schizophrenia/Schizoaffective disorder).
* Liver function tests must be within normal limits at screening.
* Participant screening for drugs with a high potential for abuse must be negative.
* Must be free of any clinically significant disease other than schizophrenia/schizoaffective disorder that would interfere with the study evaluations or procedures.
* Must have a level of understanding sufficient to communicate with research staff, cooperate with all protocol required tests and examinations, and be able to adhere to protocol restrictions and schedules.
* Must be able to understand the nature of the study and must be willing to sign an informed consent (required for each patient or the patient's authorized legal representative) prior to study enrollment.
* Females must have a follicle stimulating hormone (FSH) >=40 lU/L and be greater than 12 months since last menses or surgically sterilized.

Exclusion Criteria:

* Has a history of clinically significant local or systemic infectious disease within 4 weeks prior to initial treatment administration, clinically significant food or drug allergy, seizures, alcohol/drug dependence, previous neurosurgery, or coronary artery disease (including myocardial infarction [MI], cerebrovascular disease [stroke, transient ischemic attack (TIA)], or peripheral arterial disease).
* Has participated in a clinical trial of an investigational drug within 60 days or donated blood within the preceding 90 days prior to the start of the study.
* Has circulating human immunodeficiency virus (HIV), hepatitis C antibodies, or hepatitis B surface antigen.
* Is allergic to preladenant (SCH 420814, MK-3814) or any excipients in preladenant capsules (citric acid, lactose monohydrate, croscarmellose sodium, magnesium stearate [nonbovine, vegetable grade], Food, Drug, and Cosmetic [FD&C] blue, titanium dioxide, gelatin-national formulary [NF]).
* Females who are not surgically sterilized or postmenopausal.
* Males who are sexually active and who do not agree to use a barrier method of birth control during the study.
* Has severe/uncontrolled hypertension. (Participants with hypertension well controlled on a stable dose of standard anti-hypertensive medication for at least 4 weeks before randomization are eligible.)
* Has atrioventricular (AV) block, sick sinus syndrome, congestive heart failure, or participants with electrocardiograms (ECGs) consistent with ischemic heart disease, or significant Q waves.
* Has DSM-IV criteria of dementia (except due to schizophrenia/and schizoaffective disorder), or individuals who in the opinion of the investigator are not able to understand or comply with the study procedures or the instructions of the staff or are socially incapable to participate in the study.
* Does not comply with the requirement that participants should not use any drugs (except acetaminophen and other allowed medications) within 2 weeks prior to the study, nor alcohol (wine, beer) within 72 hours prior to drug administration.
* Judged clinically to be at suicidal risk too serious to be included in this study.
* Has received electroconvulsive therapy within 30 days before randomization.
* Is currently taking clozapine.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2006-07-10 (Actual); Primary Completion 2008-03-06 (Actual); Study Completion 2008-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/study.html?id=P04628&kw=P04628&tab=access

RESULTS

PARTICIPANT FLOW:
Period: Treatment Period 1
Arm/Group | Preladenant 25 mg BID→Placebo BID | Placebo BID→Preladenant 25 mg BID
Started | 4 | 7
Completed | 4 | 5
Not Completed | 0 | 2
Not completed — Adverse Event | 0 | 2
Period: Treatment Period 2
Arm/Group | Preladenant 25 mg BID→Placebo BID | Placebo BID→Preladenant 25 mg BID
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Preladenant 25 mg BID→Placebo BID: Participants received one preladenant 25 mg capsule BID for 14 days during the first treatment period and received one matching placebo capsule BID during the second treatment period. The 2 treatment periods were separated by a 3-week washout period.
- Total: Total of all reporting groups
Arm/Group | Preladenant 25 mg BID→Placebo BID | Placebo BID→Preladenant 25 mg BID | Total
Number analyzed (Participants) | 4 | 7 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.8 (8.5) | 46.0 (13.2) | 41.5 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Lowest Extrapyramidal Symptom Rating Score (ESRS) Total Score Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: The ESRS total score consists of 4 subscales: 1) a questionnaire of extrapyramidal symptoms (EPS) and drug-induced movement disorders (DIMD) over the previous 7 days (7 items scored as 0=Absent to 3=Severe; score range: 0-21), 2) an examination of Parkinsonism and akathisia (17 items scored as 0=None to 6=Severe; score range: 0-102), 3) an examination of dystonia (10 items scored as 0=Absent to 6=Most Severe; score range 0-60) and 4) an examination of dyskinesia (7 items scored as 0=None to 6=Severe; score range: 0-42). The ESRS total score could range from 0 to 225, with a lower score reflecting a better outcome. The lowest ESRS total score for each participant within the 6-hour range on Day 14 was analyzed.
Time Frame: Up to 6 hours post-dose on Day 14
Population: Consisted of all participants who received both treatments & had Day 14 ESRS scores from both treatment periods.
Measure: Mean (Standard Deviation); unit: Score on a scale
Groups:
- Preladenant 25 mg BID: Participants received one preladenant 25 mg capsule BID for 14 days.
- Placebo BID: Participants received one matching placebo capsule BID for 14 days.
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 11
Score on a scale
  Baseline (n=9, 11) | 14.22 (6.24) | 17.18 (11.03)
  Day 14 (n=9, 9) | 9.56 (6.64) | 10.89 (7.57)

2. Secondary Outcome: Mean ESRS Total Scores Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: The ESRS total score consists of 4 subscales: 1) a questionnaire of EPS and DIMD over the previous 7 days (7 items scored as 0=Absent to 3=Severe; score range: 0-21), 2) an examination of Parkinsonism and akathisia (17 items scored as 0=None to 6=Severe; score range: 0-102), 3) an examination of dystonia (10 items scored as 0=Absent to 6=Most Severe; score range 0-60) and 4) an examination of dyskinesia (7 items scored as 0=None to 6=Severe; score range: 0-42). The ESRS total score could range from 0 to 225, with a lower score reflecting a better outcome. The mean ESRS total scores at Hours 1, 2, 3, 4, 5, and 6 on Day 14 were analyzed.
Time Frame: 1, 2, 3, 4, 5, and 6 hours post-dose on Day 14
Population: Consisted of all participants who had a Baseline value and at least one post-Baseline value at each time point for Day 14 ESRS scores from both treatment periods. Therefore Baseline includes only participants who had corresponding data on Day 14.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 9
Score on a scale
  Baseline | 21.0 (8.6) | 20.7 (15.8)
  1 hour post-dose | 14.3 (7.0) | 15.1 (10.4)
  2 hours post-dose | 15.3 (7.1) | 13.8 (11.2)
  3 hours post-dose | 12.8 (6.6) | 14.6 (11.5)
  4 hours post-dose | 12.8 (6.7) | 14.1 (10.8)
  5 hours post-dose | 12.3 (7.0) | 13.0 (9.5)
  6 hours post-dose | 11.8 (6.7) | 11.8 (7.3)

3. Secondary Outcome: Lowest ESRS Part I Subscore: EPS and DIMD Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: The ESRS consists of 4 subscales: 1) a questionnaire of EPS and DIMD over the previous 7 days (7 items scored as 0=Absent to 3=Severe; score range: 0-21), 2) an examination of Parkinsonism and akathisia (17 items scored as 0=None to 6=Severe; score range: 0-102), 3) an examination of dystonia (10 items scored as 0=Absent to 6=Most Severe; score range 0-60) and 4) an examination of dyskinesia (7 items scored as 0=None to 6=Severe; score range: 0-42). A lower subscale score reflects a better outcome. The lowest subscale score on Day 14 was analyzed.
Time Frame: Up to 6 hours post-dose on Day 14
Population: Consisted of all participants who received both treatments & had Day 14 ESRS scores from both treatment periods.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 11
Score on a scale
  Baseline (n=9, 11) | 2.67 (1.41) | 3.00 (2.24)
  Day 14 (n=9, 9) | 1.89 (1.54) | 2.00 (1.50)

4. Secondary Outcome: Mean ESRS Part I Subscore: EPS and DIMD Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: The ESRS consists of 4 subscales: 1) a questionnaire of EPS and DIMD over the previous 7 days (7 items scored as 0=Absent to 3=Severe; score range: 0-21), 2) an examination of Parkinsonism and akathisia (17 items scored as 0=None to 6=Severe; score range: 0-102), 3) an examination of dystonia (10 items scored as 0=Absent to 6=Most Severe; score range 0-60) and 4) an examination of dyskinesia (7 items scored as 0=None to 6=Severe; score range: 0-42). A lower subscale score reflects a better outcome. The mean subscores at Hours 1, 2, 3, 4, 5 and 6 on Day 14 were analyzed.
Time Frame: 1, 2, 3, 4, 5, and 6 hours post-dose on Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 9
Score on a scale
  Baseline | 4.0 (1.9) | 4.1 (2.8)
  1 hour post-dose | 2.9 (1.8) | 2.8 (2.4)
  2 hours post-dose | 3.1 (1.8) | 2.3 (1.7)
  3 hours post-dose | 2.9 (2.0) | 2.7 (2.2)
  4 hours post-dose | 2.7 (1.9) | 2.4 (2.2)
  5 hours post-dose | 2.6 (1.7) | 2.7 (2.2)
  6 hours post-dose | 2.6 (1.7) | 2.2 (1.9)

5. Secondary Outcome: Lowest ESRS Part II Subscore: Parkinsonism and Akathisia Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: as for outcome 3
Time Frame: Up to 6 hours post-dose on Day 14
Population: Consisted of all participants who received both treatments & had Day 14 ESRS scores from both treatment periods.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 11
Score on a scale
  Baseline (n=9, 11) | 7.22 (5.04) | 8.91 (6.79)
  Day 14 (n=9, 9) | 4.67 (4.24) | 5.67 (5.74)

6. Secondary Outcome: Mean ESRS Part II Subscores: Parkinsonism and Akathisia Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: as for outcome 4
Time Frame: 1, 2, 3, 4, 5, and 6 hours post-dose on Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 9
Score on a scale
  Baseline | 10.8 (5.9) | 9.4 (5.0)
  1 hour post-dose | 8.1 (5.6) | 8.1 (6.7)
  2 hours post-dose | 9.2 (5.2) | 7.4 (8.2)
  3 hours post-dose | 7.3 (5.0) | 8.0 (7.8)
  4 hours post-dose | 7.6 (4.6) | 7.8 (7.5)
  5 hours post-dose | 7.7 (5.2) | 7.1 (6.9)
  6 hours post-dose | 6.8 (4.7) | 6.7 (6.3)

7. Secondary Outcome: Lowest ESRS Part III Subscore: Dystonia Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: as for outcome 3
Time Frame: Up to 6 hours post-dose on Day 14
Population: Consisted of all participants who received both treatments & had Day 14 ESRS scores from both treatment periods.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 11
Score on a scale
  Baseline (n=9, 11) | 1.56 (2.79) | 2.09 (4.57)
  Day 14 (n=9, 9) | 1.22 (1.99) | 1.22 (1.86)

8. Secondary Outcome: Mean ESRS Part III Subscores: Dystonia Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: as for outcome 4
Time Frame: 1, 2, 3, 4, 5, and 6 hours post-dose on Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 9
Score on a scale
  Baseline | 3.0 (4.4) | 4.2 (8.7)
  1 hour post-dose | 1.6 (2.8) | 2.2 (2.8)
  2 hours post-dose | 1.4 (2.5) | 2.0 (2.6)
  3 hours post-dose | 1.3 (2.2) | 2.1 (2.7)
  4 hours post-dose | 1.3 (2.2) | 2.0 (2.7)
  5 hours post-dose | 1.2 (2.0) | 1.8 (2.2)
  6 hours post-dose | 1.2 (2.0) | 1.3 (2.1)

9. Secondary Outcome: Lowest ESRS Part IV Subscore: Dyskinesia Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: as for outcome 3
Time Frame: Up to 6 hours post-dose on Day 14
Population: Consisted of all participants who received both treatments & had Day 14 ESRS scores from both treatment periods.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 11
Score on a scale
  Baseline (n=9, 11) | 2.00 (3.84) | 2.18 (4.12)
  Day 14 (n=9, 9) | 0.89 (2.32) | 1.22 (1.99)

10. Secondary Outcome: Mean ESRS Part IV Subscores: Dyskinesia Within the 6-hour Evaluation on Day 14 of Each Treatment Period
Description: as for outcome 4
Time Frame: 1, 2, 3, 4, 5, and 6 hours post-dose on Day 14
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Preladenant 25 mg BID | Placebo BID
Number analyzed (Participants) | 9 | 9
Score on a scale
  Baseline | 3.2 (6.4) | 2.9 (6.5)
  1 hour post-dose | 1.8 (3.6) | 2.0 (3.0)
  2 hours post-dose | 1.6 (2.9) | 2.0 (3.0)
  3 hours post-dose | 1.2 (2.6) | 1.8 (2.6)
  4 hours post-dose | 1.2 (2.6) | 1.9 (2.6)
  5 hours post-dose | 0.9 (2.3) | 1.4 (2.1)
  6 hours post-dose | 1.2 (2.6) | 1.6 (2.4)

ADVERSE EVENTS:
Time Frame: Up to 1 week after the last dose of study drug in a treatment period (Up to 8 weeks)
Description: The safety population consisted of all participants who received at least one dose of study drug. Adverse events are reported based on the study drug a participant was taking at the time of the event.
Arm/Group | Preladenant 25 mg BID | Placebo BID
Serious Adverse Events (participants affected / at risk) | 0/9 | 1/11
Other Adverse Events (participants affected / at risk) | 4/9 | 7/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 25 mg BID (N=9) | Placebo BID (N=11)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Preladenant 25 mg BID (N=9) | Placebo BID (N=11)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (4) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (2)
Feeling hot (General disorders) | 1 (1) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Crying (Psychiatric disorders) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 1 (1)
Fear (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1)
Sleep disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 1 (1)
Breast discomfort (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
This study was terminated due to low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The principal investigator agrees to provide to the sponsor 30 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the study.